CLINICAL TRIAL: NCT04731129
Title: Mini Invasive Probe Based Confocal Laser Endomicroscopy of the Pleura for Malignancies Diagnosis
Brief Title: Mini Invasive Endomicroscopy of the Pleura for Malignancies Diagnosis
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Olivier Bonhomme, Head of clinic in pulmonary medicine, University of Liege
Other Study IDs: 2018-192
Record Dates: First submitted 2020-12-22; First posted 2021-01-29 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Pleural Diseases; Pleural Neoplasms
Keywords: Probe based confocal laser endomicroscopy
MeSH Terms: conditions — Pleural Diseases; Pleural Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Probe based confocal laser endomicroscopy of the pleura — Every patient referred for medical thoracoscopy will be screened. The pCLE of the pleura will be performed 2 times. First, just before the thoracoscopy, through the Boutin's needle or the thoracentesis catheter and second through the working chanel of the pleuroscope. This last acquisition allows visual control to target the pleural endomicroscopy assessment. These two acquisitions will be compared between each other and with the histological samples of the pleuroscopy.

SUMMARY:
Recently, probe based confocal laser endomicroscopy showed to be able to distinguish malignant from benign pleura during medical thoracoscopy. However The clinical usefulness of this new tool remains to be determined.

The investigators believe that pCLE could be part of mini invasive pleural disease management and could be used during thoracentesis in order to increase the diagnostic yield of this procedure. The investigators are starting a prospective trial to recruit patients referred for medical thoracoscopy to the endoscopy unit.

First, the pCLE probe will be introduced through the Boutin's needle or the thoracentesis catheter, just before the thoracoscopy, in order to investigate the pleural pCLE features and to identify or exclude malignant infiltration. Second those features will be compared to the pCLE acquisition obtained during the medical thoracoscopy (the probe is introduced through the working chanel of the thoracoscope), under visual control. In order to compare the invasive and mini invasive acquisition, 10 criteria will be prospectively assessed.Third, These features will be compared to the histological samples performed during thoracoscopy. Finally, the interpretation of different investigators will be compared.

The 10 criteria are presented below:

1. Abnormal tissular architecture

   No: Correct identification of the previously described normal pleura characteristics Yes: identification of cellular/tissular structures which are not known to correspond to normal pleura (cellular clusters or dark clumps, glands, cells cordons, dysmorphic cells, papillar distribution….)
2. Cellular homogeneity is size, shape and fluorescence, as subjectively assessed by the investigator

   yes no
3. Mean cellular size:

   Small: < 10µm Moderate: 10 - 20µm Large: > 20µm
4. Cellular density (with reference to the Chia seed sign)

   Low (lower than the Chia seed sign) Moderate High
5. Dysplastic vessels:

   Yes: (vascular leaks, tortuous or giant vessels) No: no dysplasia
6. Vascular density (on a full optical area)

   Low: 0 -2 vessels Moderate: 3 - 4 vessels High: > 4 vessels
7. Organized or anarchic connective fibers

   Anarchic: coarse fibers, irregular in shape, without well-defined architecture Organized : regular in shape and direction, well defined architecture.
8. Chia seed sign on a full optical areal

yes No

ELIGIBILITY:
Inclusion Criteria:

* Every patient referred to the endoscopy unit for medical thoracoscopy

Exclusion Criteria:

* Pregnancy
* Known allergy to the fluorescein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient referred to the endoscopy unit for medical thoracoscopy
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duysinx Bernard, PhD, Study Director — University of Liege
Locations (1):
- Olivier Bonhomme, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Referred to Medical Throacoscopy for Treatment or Exploration of a Pleural Effusion: Every patient referred to medical thoracoscopy for pleural effusion treatment or workup. exclusion criteria are age< 18; Pregnancy; Known allergy to fluorescein
Period: Overall Study
Arm/Group | Patients Referred to Medical Throacoscopy for Treatment or Exploration of a Pleural Effusion
Started | 59
Completed | 52
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Patients Referred to Medical Throacoscopy for Treatment or Exploration of a Pleural Effusion
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 8 patients unwilling to participate
  years | 67 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 52

OUTCOME MEASURES:

1. Primary Outcome: Malignant Pleural Infiltration Identification
Description: Before medical thoracoscopy, the laser endomicroscopy probe will be introduced through the Boutin's needle or the thoracentesis catheter. The pleural probe based confocal laser endomicroscopy acquisition will be assessed by two experienced and unblinded clinicians (aware of the medical history of the patient) during the procedure. The objective is to determine if the preselected criteria are present with significantly different frequencies in malignant adn in benign pleural involvement.
Time Frame: one day
Measure: Count of Participants; unit: Participants
Groups:
- Patietns With a Pleural Biopsy Histology of Benign Disease: Every patients had pleural biopsies to conclude the thoracoscopy. This group gather patients with a benign pleural effusion according to pleural biopsies
- Patients With a Malignant Pleural Biopsy Histology: Every patient included had pleural biopsies at the end of the medical thoracoscopy. This group gathers patients with a malignant pleural effusion according to pleural biopsies.
Arm/Group | Patietns With a Pleural Biopsy Histology of Benign Disease | Patients With a Malignant Pleural Biopsy Histology
Number analyzed (Participants) | 21 | 31
Participants
  Abnormal tissular architecture: Yes | 12 | 27
  Abnormal tissular architecture: No | 9 | 4
  Homogeneous cell size: Yes | 15 | 10
  Homogeneous cell size: No | 6 | 21
  Homogeneous cell shape: Yes | 15 | 10
  Homogeneous cell shape: No | 6 | 21
  Homogeneous cell fluorescence: Yes | 11 | 7
  Homogeneous cell fluorescence: No | 10 | 24
  Blood vessel dysplasia: Yes | 9 | 20
  Blood vessel dysplasia: No | 12 | 11
  Organized conjunctive fibers: Yes | 19 | 23
  Organized conjunctive fibers: No | 2 | 8
  Full Chia seed sign: Yes | 6 | 2
  Full Chia seed sign: No | 15 | 29
  General physician conclusion: Yes | 10 | 27
  General physician conclusion: No | 11 | 4
Statistical Analysis 1: Comparison: Patietns With a Pleural Biopsy Histology of Benign Disease vs Patients With a Malignant Pleural Biopsy Histology; Abnormal tissular architecture; Test type: Superiority; p = 0.023, Fisher Exact — threshold for statistical significance < 0.05
Statistical Analysis 2: Comparison: Patietns With a Pleural Biopsy Histology of Benign Disease vs Patients With a Malignant Pleural Biopsy Histology; Homogeneous cell size; Test type: Superiority; p = 0.01, Fisher Exact — Threshold for statistical significance < 0.05
Statistical Analysis 3: Comparison: Patietns With a Pleural Biopsy Histology of Benign Disease vs Patients With a Malignant Pleural Biopsy Histology; Homogeneous cell shape; Test type: Superiority; p = 0.01, Fisher Exact — threshold for statistical significance < 0.05
Statistical Analysis 4: Comparison: Patietns With a Pleural Biopsy Histology of Benign Disease vs Patients With a Malignant Pleural Biopsy Histology; Homogeneous cell fluorescence; Test type: Superiority; p = 0.013, Fisher Exact — threshold for statistical significance < 0.05
Statistical Analysis 5: Comparison: Patietns With a Pleural Biopsy Histology of Benign Disease vs Patients With a Malignant Pleural Biopsy Histology; Blood vessel dysplasia; Test type: Superiority; p = 0.16, Fisher Exact — threshold for statistical significance < 0.05
Statistical Analysis 6: Comparison: Patietns With a Pleural Biopsy Histology of Benign Disease vs Patients With a Malignant Pleural Biopsy Histology; Organized conjunctive fibers; Test type: Superiority; p = 0.17, Fisher Exact — threshold for statistical significance < 0.05
Statistical Analysis 7: Comparison: Patietns With a Pleural Biopsy Histology of Benign Disease vs Patients With a Malignant Pleural Biopsy Histology; Full chia seed sign; Test type: Superiority; p = 0.049, Fisher Exact — threshold for statistical significance < 0.05
Statistical Analysis 8: Comparison: Patietns With a Pleural Biopsy Histology of Benign Disease vs Patients With a Malignant Pleural Biopsy Histology; General physician conclusion; Test type: Superiority; p = 0.0041, Fisher Exact — threshold for statistical significance < 0.05

2. Primary Outcome: Concordance Between the Mini Invasive Assessment and the Invasive Pleural Assessment.
Description: Every (Serious)adverse event will be reported during the intervention or during post intervention surveillance (1 hour post intervention).
  The feasibility will be assessed by comparing the images from the mini invasive phase with this from the invasive phase.
Time Frame: One day
Measure: Count of Participants; unit: Participants
Groups:
- The Entire Studied Population: Every patient included had pleural biopsies at the end of the medical thoracoscopy.
Arm/Group | The Entire Studied Population
Number analyzed (Participants) | 52
Participants
  Abnormal tissular architecture: concordant | 49
  Abnormal tissular architecture: non concordant | 3
  Homogeneous cell shape: concordant | 50
  Homogeneous cell shape: non concordant | 2
  Homogeneous cell fluorescence: concordant | 50
  Homogeneous cell fluorescence: non concordant | 2
  Homogeneous cell size: concordant | 50
  Homogeneous cell size: non concordant | 2
  Full chia seed sign: concordant | 52
  Full chia seed sign: non concordant | 0
  General physician conclusion: concordant | 52
  General physician conclusion: non concordant | 0

3. Primary Outcome: Pleural Fluid Cytological Analysis
Description: Pathological analysis of the collected pleural fluid is compared to the final histological diagnosis of pleural biopsies.
Time Frame: one day
Measure: Count of Participants; unit: Participants
Arm/Group | Patietns With a Pleural Biopsy Histology of Benign Disease | Patients With a Malignant Pleural Biopsy Histology
Number analyzed (Participants) | 21 | 31
Participants
  Benign fluid cytology | 21 | 18
  malignant pleural fluid cytology | 0 | 13

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | The Entire Studied Population
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04731129/Prot_SAP_002.pdf
  • Informed Consent Form (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT04731129/ICF_001.pdf